CLINICAL TRIAL: NCT06938165
Title: The Safety and Efficacy of Fecal Microbiota Transplant for Steroid-refractory Graft-versus-host Disease
Brief Title: The Safety and Efficacy of Fecal Microbiota Transplant (FMT) for Steroid-refractory Graft-versus-host Disease
Acronym: FMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2020-194
Record Dates: First submitted 2025-04-10; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: GVHD
Keywords: GVHD
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with refractory graft-versus-host disease (Experimental): FMT for patients with refractory GVHD
  Interventions: Other: Fecal Microbiota Transplant (FMT)

INTERVENTIONS:
Other: Fecal Microbiota Transplant (FMT) — FMT in patients with refractory GVHD

SUMMARY:
This clinical study evaluates the safety and efficacy of fecal microbiota transplantation (FMT) in patients with steroid-refractory graft-versus-host disease (GVHD).

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to sign the informed consent form and complete follow-up;
2. Aged 18-65 years, regardless of gender;
3. Patients with refractory GVHD.

Exclusion Criteria:

1. life-threatening or associated with severe non-GvHD complications;
2. Persistent malignant conditions;
3. Patients who have undergone second or multiple hematopoietic stem cell transplants;
4. History of severe allergic reactions;
5. Any condition that the investigator considers unsuitable for inclusion (such as any history, treatment history, or abnormal test data that may confound the study results, interfere with full participation in the study, or harm the patient's interests);

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 12 weeks
  Assessment of ORR (ORR = Complete Response (CR) + Partial Response (PR)) at 12 weeks after treatment. CR was defined as the complete resolution of all disease manifestations in every affected organ or site. PR was defined as an improvement in at least one organ or site without any disease progression occurring in other organs or sites.

SECONDARY OUTCOMES:
Number of Participants Experiencing an Adverse Event (AE) | 12 weeks
  An adverse event refers to any unfavorable and unintended sign, symptom, or illness temporally associated with the use of the product, regardless of whether it is considered related to the product. A serious adverse event (SAE) is defined as an AE that results in death, is life-threatening, causes persistent or significant disability/incapacity, necessitates or extends hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Only accept academic purpose for the sharing data and please contact PI with reasonable inquiring.

REFERENCES:
- [Derived] Yang K, Du J, Huang F, Si Y, Gu Y, Xu N, Fan Z, Xue R, Wang P, Yao X, Liu H, Li X, Xu J, Wang Z, Sun J, Chen Y, Xuan L, Liu Q. Fecal microbiota transplantation for refractory chronic graft-versus-host disease after allogeneic hematopoietic cell transplantation: a pilot open-label, non-placebo-controlled study. BMC Med. 2025 Aug 26;23(1):498. doi: 10.1186/s12916-025-04336-z. PMID 40859356